CLINICAL TRIAL: NCT05319236
Title: A Prospective, Multicentric Interventional Study Assessing the Range of Most Clinically Relevant Indications for Use of the Non-invasive Wireless Gabi System for the Recording, in Non-motion Condition, of SpO2, Pulse Rate, Respiratory Rate and Movements of Young Children With Underlying Medical Conditions.
Brief Title: Clinical Use Cases Assessment of the Gabi System in Young Children With Underlying Medical Conditions (BRIDGE Study)
Acronym: BRIDGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gabi SmartCare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: R-DND-11 BRIDGE Study_CIP
Record Dates: First submitted 2022-03-22; First posted 2022-04-08 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-02

CONDITIONS: Cardiac Disease; Respiratory Disease; Congenital Cardiac Defect; Cardiovascular Diseases; Chronic Respiratory Disease; Chronic Cardiopulmonary Disease; Premature Infant Disease
MeSH Terms: conditions — Heart Diseases; Respiration Disorders; Heart Defects, Congenital; Cardiovascular Diseases; Pulmonary Heart Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Gabi System (Other): Subjects will wear the Gabi system each time they go to sleep or are resting, to measure and record their SpO2, pulse rate, respiratory rate and movements.
  Interventions: Device: Gabi System

INTERVENTIONS:
Device: Gabi System — See arm description

SUMMARY:
Subjects will use the Gabi system on a daily basis for 3 months, each time the subject is resting or asleep. The Gabi system will recording the SpO2, pulse rate, respiratory rate and movements of the subject.

The objective of this study is to perform a first assessment of the range of most potentially clinically relevant indications for use of the Gabi system for children < 6 years old with underlying medical conditions.

This is performed by asking HCPs to review the data measured by the Gabi system after taking a medical decision independently from the Gabi data and to assess the potential clinical utility of the Gabi system.

The usability of the system will also be assessed throughout questionnaires filled out by the HCPs and by the caregivers.

*During this study, the data collected by the Gabi system are not intended to be used by caregivers or HCPs to take any (medical) decisions.

ELIGIBILITY:
Inclusion Criteria:

1. Infants and children < 6 years old.
2. Subjects who present at least one of the following underlying medical conditions:

   1. Subjects who underwent a congenital cardiac or cardiopulmonary surgery recently and could benefit from an additional post-surgery monitoring at home, per the investigator's opinion.
   2. Subjects at risk awaiting surgery.
   3. Subjects hospitalized following a severe respiratory condition within the past 2 weeks requiring invasive or non-invasive ventilation or oxygen therapy.
   4. Subjects hospitalized following a severe cardiovascular condition within the past 2 weeks, including severe heart failure, tachycardia or bradycardia.
   5. Subjects with chronic respiratory disease, such as asthma, developmental or cardiovascular conditions who could benefit from medical monitoring at home, per the investigator's opinion.
   6. Subjects with chronic respiratory support at home.
   7. Premature babies who required intensive neonatal care.
   8. Subjects hospitalized following a Brief Resolved Unexpected Event (BRUE) within the past 2 weeks.
   9. A clinical risk identified by the investigator which justifies the potential benefit of having a Gabi system used by the subject
3. Subject is (or is willing to be) followed up by an HCP of the investigation site during the duration of the study.
4. Signed informed consent form prior to performing any study specific procedure.
5. Willing and likely (based on the investigator's judgement) to comply with all study requirements.

Exclusion Criteria:

1. Weight < 2.5 kg.
2. Subject presenting an anatomical limitation that would prevent the use of the Gabi system.
3. Subjects presenting a motor disorder that would prevent the use of the Gabi system (with the exception of epilepsy ).
4. Subjects participating in another interventional clinical study (with the exception of registries), which may have an impact on this study outcomes, based on the investigator's judgement.

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2022-02-16 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Clinical Utility | Assessed at the end of the 3-month period for each participant
  Define the range of most potentially clinically significant indications for use of the Gabi system based on the Gabi system clinical utility assessment per medical condition, assessed throughout Medical Decision Questionnaires and Clinical Utility Questionnaires.
Caregiver Usability | Assessed at the end of the 3-month period for each participant
  Assess the usability of the Gabi system from the point of view of the caregivers through a Usability Questionnaire.
HCP Usability | Assessed at the end of the 3-month period for each participant
  Assess the usability of the Gabi system from the point of view of the HCPs through a Usability Questionnaire.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (2):
  - Children's National Hospital, Washington D.C., District of Columbia
  - Columbia University Irving Medical Center, New York, New York
- Belgium (2):
  - Universitair Ziekenhuis Antwerpen (UZA), Antwerp
  - Clinique CHC Montlégia, Liège

IPD SHARING:
Plan to Share IPD: No